CLINICAL TRIAL: NCT04780269
Title: Foley Catheter Versus Prostaglandin E2 Vaginal Suppository for Labor Induction at Term: a Pilot Study
Brief Title: Foley Catheter Versus PGE2 for Labor Induction at Term: a Pilot Study
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: understaffed
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Zehong Zhou, Principle investigator, Guangzhou Women and Children's Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: [2020]31201
Record Dates: First submitted 2021-02-22; First posted 2021-03-03 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Labor Induction; Induced Delivery
Keywords: Labor induction; Term delivery with an unfavorable cervix; Foley catheter; Prostaglandin E2
MeSH Terms: interventions — Labor, Induced; Dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Induction of labor with Foley catheter (Experimental): A Foley catheter will be introduced transcervically in women allocated in this group.
  Interventions: Device: Induction of labor with Foley catheter
- Induction of labor with PGE2 (Experimental): PGE2 (1mg) will be inserted into the posterior vaginal fornix.
  Interventions: Drug: Induction of labor with PGE2

INTERVENTIONS:
Device: Induction of labor with Foley catheter — A Foley catheter will be introduced transcervically in women allocated in this group, with the aid of a vaginal speculum after cervical cleaning with an aseptic solution. The balloon will be inflated with 60 mL of sterile 0.9%% sodium chloride (NaCl) after insertion past the internal os. The external end of the catheter is taped to the inner thigh without applying any traction or tension.
  Other Names: Foley Catheter
  Arms: Induction of labor with Foley catheter
Drug: Induction of labor with PGE2 — PGE2 (1mg) will be inserted into the posterior vaginal fornix. Women will be assigned one hour of bed rest while continuously monitored by cardiotocography.
  Other Names: Dinoprostone suppositories
  Arms: Induction of labor with PGE2

SUMMARY:
Induction of labor is one of the most common interventions in obstetrics. In the past decade, the rates of labor induction at term have doubled from approximately 9% to 23% in the United States and from 10% to 20.4% in China. The majority of women undergoing labor induction requires cervical ripening for the unfavorable cervixes. As globally, it is still required to explore an optimal induction method. Foley catheter was among the oldest mechanical approaches, while prostaglandin E2 vaginal suppository (PGE2) one of the most popular pharmacological agents for cervical ripening. There were studies reporting similar cesarean section rates between these two methods. However, there are no randomized control trials (RCTs) with adequate power to compare their frequencies of severe perinatal complications. The investigators aim to compare the effectiveness and safety of Foley catheter versus PGE2 for induction of labor among term pregnant women with an unfavourable cervix.

DETAILED DESCRIPTION:
The investigators propose a single center, open-label, randomized controlled clinical trial (1:1 treatment ratio) in Guangzhou Women and Children's Medical Center. Women with a term pregnancy, an indication for induction of labor, and a live singleton fetus at cephalic presentation, intact membranes, an unfavorable cervix, no prior cesarean section or contraindication to vaginal delivery, are eligible to participate. After informed consent, they will be randomized to undergo induction of labor by Foley catheter or PGE2.

Our primary outcomes will be (I) a composite of severe perinatal complications and (II) vaginal delivery. Before the formal recruitment of this RCT, a pilot study with a sample size of 200 pregnant women will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Women scheduled for induction of labor.
* Women aged ≥ 18 years old
* ≥ 37 weeks of gestation
* Live singleton pregnancy in cephalic presentation
* Intact membranes
* Cervical Bishop score < 6
* Informed consent.

Exclusion Criteria:

* Contraindications for vaginal delivery.
* Prior cesarean section
* Known hypersensitivity for Foley catheter or PGE2
* Non-reassuring fetal status
* Lethal fetal congenital anomaly

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of cases with perinatal complications | Up to 3 weeks
  This primary outcome will be a composite of cases with severe perinatal complications and consists of one or more of the following: need for respiratory support within hours after birth, Apgar score < 7 at 1 minutes, Apgar score <7 at 5 minutes, umbilical cord arterial potential of hydrogen (pH ) < 7.10, birth trauma (including bone fracture, neurologic injury, or retinal hemorrhage), hypoxic-ischemic encephalopathy or need for therapeutic hypothermia, seizure, pneumonia, meconium aspiration syndrome, neonatal meningitis, neonatal sepsis, infant respiratory distress syndrome, pneumothorax or pneumomediastinum, apnoea, necrotising enterocolitis, clinical diagnosis of asphyxia, intraventricular haemorrhage, perinatal death (fetal or neonatal death occurring during childbirth, or up to 7 completed days after birth) or admission to the neonatal intensive care unit (NICU) for >48 hours. Each component of this outcome is described from outcome 3 to outcome 21.
Percentage of vaginal delivery | Up to 1 week
  The co-primary outcome is vaginal delivery.

SECONDARY OUTCOMES:
Number of neonates need for respiratory support | Up to 1 week
  Respiratory support within hours after birth
Number of neonates with Apgar score < 7 at 1 minutes | On the day of delivery
  Apgar scores of less than 7 at 1 min
Number of neonates with Apgar score < 7 at 5 minutes | On the day of delivery
  Apgar scores of less than 7 at 5 min
Number of neonates with umbilical cord arterial pH < 7.10 | On the day of delivery
  An assay of arterial cord blood pH of less than 7.10
Number of neonates with birth trauma | Up to 1 week
  Birth trama including bone fracture, neurologic injury, or retinal hemorrhage
Number of neonates with hypoxic-ischemic encephalopathy or need for therapeutic hypothermia | Up to 1 week
  Neonates diagnosed with hypoxic-ischemic encephalopathy or require therapeutic hypothermia
Number of neonates with pneumonia | Up to 2 weeks
  Pneumonia revealed by physical examination, blood test and image
Number of neonates with seizure | Up to 2 weeks
  Clinical signs of seizure
Number of neonates with meconium aspiration syndrome | Up to 2 week
  Diagnosed according to clinical symptoms, blood test and image
Number of neonates with neonatal meningitis | Up to 4 weeks
  Diagnosed by blood and cerebrospinal fluid test and image
Number of neonates with neonatal sepsis | Up to 2 weeks
  Diagnosed by clinical symptoms, blood test and bacterial culture
Number of neonates with infant respiratory distress syndrome | Up to 2 weeks
  Diagnosed by blood test and image
Number of neonates with infant pneumothorax or pneumomediastinum | Up to 2 weeks
  Diagnosed by thorax image
Number of neonates with apnoea | Up to 2 weeks
  Clinical diagnosis of apnoea
Number of neonates with necrotising enterocolitis | Up to 2 weeks
  Diagnosed by clinical symptoms, stool examination and image
Number of neonates with clinical diagnosis of asphyxia | Up to 2 weeks
  Clinical diagnosis of neonatal asphyxia
Number of perinatal deaths | up to 2 weeks
  Fetal or neonatal death occurring during childbirth
Number of neonates with intraventricular hemorrhage | Up to 2 week
  Intraventricular haemorrhage diagnosed by clinical symptoms and image
Number of neonates admission to the NICU for >48 hours | up to 2 weeks
  Length of admission to the NICU for less than 48 hours
Number of cases with maternal secondary outcomes | Up to 2 weeks
  This secondary outcome will be a composite of maternal complications and consists of one or more of the following: cardio-respiratory arrest, damage to internal organs (bowel, bladder or ureters), postpartum hemorrhage (estimated blood loss >500 milliliter (mL) in the 24 hours after delivery), hysterectomy for any complications resulting from birth, intensive care admission, uterine rupture: separation of the uterine wall, maternal infection, pulmonary embolism, stroke, maternal satisfaction, maternal death. Each component of this outcome is described from outcome 23 to outcome 33.
Number of mothers with cardio-respiratory arrest | Up to 2 weeks
  Clinical diagnosis of cardio-respiratory arrest
Number of mothers with damage to internal organs | Up to 2 weeks
  Damage to internal organs, including bowel, bladder or ureters
Number of mothers with postpartum hemorrhage | Up to 1 week
  Postpartum hemorrhage is defined as estimated blood loss >500 mL in the 24 hours after delivery
Number of mothers have hysterectomy | Up to 2 weeks
  Hysterectomy for any complications resulting from birth
Number of mothers have intensive care admission | Up to 3 weeks
  Admission of puerpera to ICU
Number of mothers have uterine rupture | Up to 2 weeks
  Uterine rupture refers to separation of the uterine wall
Number of maternal infection | Up to 2 weeks
  Maternal infection diagnosed by clinical symptoms, blood test, bacterial culture.
Number of mothers have pulmonary embolism | Up to 2 weeks
  Diagnosed by clinical symptoms, blood test and image
Number of mothers have stroke | Up to 2 weeks
  Diagnosed by clinical signs, blood test and cerebral image
Scores of maternal satisfaction with the intervention of labor induction | Up to 2 weeks
  Maternal satisfaction will be evaluated by a questionaire consisted of 11 questions scored on a 5-point Likert scale.
Number of maternal death | Up to 2 weeks
  Maternal death due to delivery
Number of neonates with hyperbilirubinemia | Up to 2 weeks
  Hyperbilirubinemia requiring photo-therapy or exchange transfusion
Number of neonates with hypoglycemia | Up to 2 weeks
  Hypoglycemia requiring intravenous therapy
Length of neonatal admission (days) | Up to 3 weeks
  Length of admission of neonate
Number of neonates with cephalohematoma | Up to 2 weeks
  Diagnosed by physical examination and image
Number of neonates have shoulder dystocia | Up to 1 week
  Diagnosed by physical examination and image
Number of neonates have admission to the NICU < 48 hours | Up to 1 week
  Admission of neonates to NICU for less than 48 hours
Number of cases with indication of caesarean section | Up to 1 week
  Indication of caesarean section including failure to progress at first stage, failure to progress at second stage, failed instrumental delivery, suspected fetal distress, suspected fetal distress and failure to progress at first stage, suspected fetal distress and failure to progress at second stage, and maternal complications or other
Number of cases with indication of instrumental delivery | Up to 1 week
  Indication of instrumental delivery including failure to progress at second stage, suspected fetal distress, suspected fetal distress and failure to progress at second stage, and maternal complications or other

OTHER OUTCOMES:
Number of cases with suspected intrapartum infection | Up to 1 week
  Temperature ≥ 38°C during labor and/or use of broad-spectrum antibiotics due to suspected infection
Number of cases with uterine hyperstimulation | Up to 1 week
  Single contractions lasting 2 minutes or more, or five or more contractions in a 10 minutes period more than one induction agent required

CONTACTS AND LOCATIONS:
Overall Officials: JinYing Yang, MD., Principal Investigator — Guangzhou Women and Children's Medical Center
Locations (1):
- Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin JA, Hamilton BE, Sutton PD, Ventura SJ, Mathews TJ, Osterman MJ. Births: final data for 2008. Natl Vital Stat Rep. 2010 Dec 8;59(1):1, 3-71. PMID 22145497
- [Background] Grobman WA, Rice MM, Reddy UM, Tita ATN, Silver RM, Mallett G, Hill K, Thom EA, El-Sayed YY, Perez-Delboy A, Rouse DJ, Saade GR, Boggess KA, Chauhan SP, Iams JD, Chien EK, Casey BM, Gibbs RS, Srinivas SK, Swamy GK, Simhan HN, Macones GA; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Labor Induction versus Expectant Management in Low-Risk Nulliparous Women. N Engl J Med. 2018 Aug 9;379(6):513-523. doi: 10.1056/NEJMoa1800566. PMID 30089070
- [Background] Jozwiak M, Oude Rengerink K, Benthem M, van Beek E, Dijksterhuis MG, de Graaf IM, van Huizen ME, Oudijk MA, Papatsonis DN, Perquin DA, Porath M, van der Post JA, Rijnders RJ, Scheepers HC, Spaanderman ME, van Pampus MG, de Leeuw JW, Mol BW, Bloemenkamp KW; PROBAAT Study Group. Foley catheter versus vaginal prostaglandin E2 gel for induction of labour at term (PROBAAT trial): an open-label, randomised controlled trial. Lancet. 2011 Dec 17;378(9809):2095-103. doi: 10.1016/S0140-6736(11)61484-0. Epub 2011 Oct 24. PMID 22030144
- [Background] Saad AF, Villarreal J, Eid J, Spencer N, Ellis V, Hankins GD, Saade GR. A randomized controlled trial of Dilapan-S vs Foley balloon for preinduction cervical ripening (DILAFOL trial). Am J Obstet Gynecol. 2019 Mar;220(3):275.e1-275.e9. doi: 10.1016/j.ajog.2019.01.008. Epub 2019 Feb 18. PMID 30790569
- [Background] Dos Santos F, Drymiotou S, Antequera Martin A, Mol BW, Gale C, Devane D, Van't Hooft J, Johnson MJ, Hogg M, Thangaratinam S. Development of a core outcome set for trials on induction of labour: an international multistakeholder Delphi study. BJOG. 2018 Dec;125(13):1673-1680. doi: 10.1111/1471-0528.15397. Epub 2018 Sep 10. PMID 29981523
- [Background] Ten Eikelder ML, Oude Rengerink K, Jozwiak M, de Leeuw JW, de Graaf IM, van Pampus MG, Holswilder M, Oudijk MA, van Baaren GJ, Pernet PJ, Bax C, van Unnik GA, Martens G, Porath M, van Vliet H, Rijnders RJ, Feitsma AH, Roumen FJ, van Loon AJ, Versendaal H, Weinans MJ, Woiski M, van Beek E, Hermsen B, Mol BW, Bloemenkamp KW. Induction of labour at term with oral misoprostol versus a Foley catheter (PROBAAT-II): a multicentre randomised controlled non-inferiority trial. Lancet. 2016 Apr 16;387(10028):1619-28. doi: 10.1016/S0140-6736(16)00084-2. Epub 2016 Feb 3. PMID 26850983